CLINICAL TRIAL: NCT04919070
Title: 'Connect for Caregivers' - Developing a Brief Intervention for Social Connectedness
Brief Title: Connect for Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sally Norton, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00004316; P30AG064103 (NIH)
Record Dates: First submitted 2021-06-02; First posted 2021-06-09 (Actual); Results first posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Social Isolation; Loneliness
Keywords: Social Connectedness
MeSH Terms: conditions — Social Isolation | interventions — Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Connect for Caregivers (Experimental): Connect for Caregivers is a single session behavioral intervention with three components: 1) psychoeducation on the importance of connectedness for health and well-being; a card sort-based discussion prioritization tool that systematizes and routinizes the process of identifying and prioritizing barriers to connectedness; 3) personalized resources to address the identified barriers and targets.
  Interventions: Behavioral: Connect for Caregivers

INTERVENTIONS:
Behavioral: Connect for Caregivers — The intervention being studied is a single session guided behavioral intervention to improve social connectedness in caregivers of individuals with ADRD. The intervention, Connect for Caregivers, provides psychoeducation on the importance of social connectedness for health and well-being, includes a card-sort process to identify and prioritize barriers to connectedness, and provides personalized resources and strategies for caregivers to use to increase their social connectedness.

SUMMARY:
Connect for Caregivers is a intervention feasibility pilot study. The purpose of the study is to pilot test a newly developed single session behavioral intervention to help caregivers of individuals with Alzheimer's Disease or related dementias gain understanding of the importance of increasing social connectedness, awareness of their personal barriers to connectedness, and knowledge of local resources for promoting connectedness.

DETAILED DESCRIPTION:
Connect for Caregivers is a intervention feasibility pilot study. We use a mixed methods approach to initiate the development and testing process for a single session behavioral intervention to help caregivers gain understanding of the importance of increasing connectedness, awareness of their personal barriers to connectedness, and knowledge of local resources for promoting connectedness. The intervention-"Connect 4 Caregivers"-has three components: 1) psychoeducational materials on the importance of connectedness for health and wellbeing; 2) a card sort-based 'discussion prioritization tool' that systematizes and routinizes the process of identifying and prioritizing barriers to connectedness; 3) personalized resources to address the identified barriers/targets.

Aim 1 is to investigate whether Connect for Caregivers is associated with a signal for efficacy for changing connectedness by having n=5 caregivers complete the single session intervention and provide quantitative and qualitative data on their experience with the intervention and motivation to work on increasing their social connectedness (a signal for potential efficacy).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 yrs;
2. English speaking;
3. Caregiver (age 50 or older) for a community-dwelling family member with ADRD, living with (or in close proximity to) family member with dementia;
4. Elevated caregiving distress: Above population mean (>11) on 10-item Perceived Stress Scale (PSS-10) and/or at least moderate caregiver strain (score >= 5) on the Modified Caregiver Strain Index (MCSI).
5. Social connectedness: UCLA Loneliness Scale: Short Form score of >5.

Exclusion Criteria:

1. Primary language is not English;
2. Current problem drinking on the AUDIT-C (score of 5 or greater indicating exclusion);
3. Current non-alcohol psychoactive substance abuse (MINI Neuropsychiatric Interview), psychotic disorders (current and lifetime, MINI), bipolar disorder (MINI), and current mood disorder with psychotic features (MINI);
4. Significant cognitive impairment (MOCA <22); and
5. Hearing problems that preclude completion of the intervention.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include self-reported demographic data from interviews with 5 older adults who are caregivers for individuals with ADRD. Data from this research will be made available to the public in the University of Rochester's institutional repository, UR Research, at https://urresearch.rochester.edu. We will share the research protocols, in a text format, such as MS Word or PDF. For quantitative data, the PI will make available the actual datasets generated from research, in a commonly- used format such as a SAS® dataset. The datasets will be associated with a related publication, research protocol or other documentation of the original research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Timetable to release the data: the data and referenced resources from publications will be made available by the on-line publication date.
Access Criteria: The investigators will make the data and associated documentation available to users only under a data-sharing agreement as suggested by the NIH that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. 4. De-identification of data from human subjects: A final complete database will be created to host all data which will be stripped of any identifiers and stored pursuant to UR Institutional Review Board protocols.
URL: https://urresearch.rochester.edu

REFERENCES:
- [Derived] Norton SA, Carter RM, Moskow M, Bobry M, Wittink MN, Heffner KL, Van Orden KA. Connect for caregivers: an exemplar using the NIH Stage Model for behavioral intervention development. Aging Ment Health. 2025 Nov 6:1-11. doi: 10.1080/13607863.2025.2581098. Online ahead of print. PMID 41196573

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Connect for Caregivers
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Caregivers of a family member with dementia.
Arm/Group | Connect for Caregivers
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.89 (4.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Perceived Autonomy [Mean (Standard Deviation); unit: score on a scale] — This is a self-report measure that assesses a mechanism posited by Self-Determination Theory to increase motivation for healthy behaviors. It has 6 items, a range from 6-30, and higher scores indicate greater perceived autonomy.
  score on a scale | 21.8 (1.66)
Perceived Competence [Mean (Standard Deviation); unit: score on a scale] — This is a self-report measure that assesses a mechanism posited by Self-Determination Theory to increase motivation for healthy behaviors. It has 7 items, a range from 7-35, and higher scores indicate greater perceived competence.
  score on a scale | 16.8 (1.28)
Knowledge of Social Engagement [Mean (Standard Deviation); unit: score on a scale] — This is a self-report measure that assesses a subject's knowledge of the importance of social connections. It has 4 items, a range from 4-20, and higher scores indicate greater knowledge.
  score on a scale | 14.8 (2.59)
UCLA Loneliness Scale [Mean (Standard Deviation); unit: score on a scale] — UCLA Loneliness Scale Version 3, which assesses self-reported loneliness. 20 items, rated as to how often the participant has felt a certain way in the prior month (e.g., "How often do you feel alone?") -- "never" (1), "rarely" (2), "sometimes" (3), or "often" (4). Higher scores indicate greater loneliness. Total scores range from 20 to 80, with higher scores representing a worse outcome (i.e., greater loneliness).
  score on a scale | 49.6 (10.85)

OUTCOME MEASURES:

1. Primary Outcome: Perceived Autonomy
Description: This is a self-report measure that assesses a mechanism posited by Self-Determination Theory to increase motivation for healthy behaviors. It has 6 items, a range from 6-30, and higher scores indicate greater perceived autonomy.
Time Frame: two weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect for Caregivers
Number analyzed (Participants) | 5
score on a scale | 21.2 (1.32)

2. Primary Outcome: Perceived Competence Scale
Description: This is a self-report measure that assesses a mechanism posited by Self-Determination Theory to increase motivation for healthy behaviors. It has 7 items, a range from 7-35, and higher scores indicate greater perceived competence.
Time Frame: two weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect for Caregivers
Number analyzed (Participants) | 5
score on a scale | 16.4 (2)

3. Secondary Outcome: Knowledge of Social Engagement
Description: This is a self-report measure that assesses a subject's knowledge of the importance of social connections. It has 4 items, a range from 4-20, and higher scores indicate greater knowledge.
Time Frame: two weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect for Caregivers
Number analyzed (Participants) | 5
score on a scale | 15.6 (2.3)

4. Secondary Outcome: Loneliness
Description: UCLA Loneliness Scale Version 3, which assesses self-reported loneliness. 20 items, rated as to how often the participant has felt a certain way in the prior month (e.g., "How often do you feel alone?") -- "never" (1), "rarely" (2), "sometimes" (3), or "often" (4). Higher scores indicate greater loneliness. Total scores range from 20 to 80, with higher scores representing a worse outcome (i.e., greater loneliness).
Time Frame: two weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect for Caregivers
Number analyzed (Participants) | 5
score on a scale | 53.4 (6.11)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Connect for Caregivers
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT04919070/Prot_SAP_000.pdf